CLINICAL TRIAL: NCT05684692
Title: Screening Trial for Pain Relief in Schwannomatosis (STARFISH)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); RECORDATI GROUP (Industry)
Responsible Party: Principal Investigator, Scott R. Plotkin, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-512
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Schwannomatosis; Schwannomas; Pain, Chronic
Keywords: Schwannomatosis; Schwannomas; Pain; chronic Pain; Severe Pain
MeSH Terms: conditions — Schwannomatosis; Neurilemmoma; Chronic Pain; Pain | interventions — siltuximab; erenumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: (1) Double-Blind period for Siltuximab or Placebo Arm; and (2) Single-Blind period for Erenumab-Aooe or Placebo Arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sub-study A: Siltuximab (Experimental): The treatment period includes a double-blind treatment period (days 1-84) and an open-label treatment period (days 85-168).
  All participants will receive siltuximab during this drug sub-study. Twenty (20) participants will be randomized to receive either Siltuximab or matching placebo during the double-blind treatment period. All participants will receive siltuximab during the open-label treatment period. Participants will complete study procedures as outlined:
  * Double-Blind Treatment period: Administration of Siltuximab versus matching placebo in pre-determined dose once every 21 days (for 4 cycles).
  * Open-Label Treatment period: Administration of Siltuximab in pre-determined dose once every 21 days (for 4 cycles).
  Interventions: Drug: Siltuximab; Drug: Siltuximab Matching Placebo
- Sub-study B: Erenumab-Aooe (Experimental): The treatment period includes a single-blind treatment period (days 1-84) and an open-label treatment period (days 85-168).
  All participants will receive erenumab-aooe during this drug sub-study. Twenty (20) participants will receive a randomization assignment to receive either Erenumab-Aooe or matching placebo during the single-blind treatment period. All participants will receive erenumab-aooe during the open-label treatment period. Participants will complete study procedures as outlined:
  * Single-Blind treatment period (days 1 - 84): Administration of Erenumab-Aooe versus matching placebo in pre-determined dose once every 28 days (for 3 cycles).
  * Open-Label Treatment period (days 85-168): Administration of Erenumab-Aooe in pre-determined dose once every 28 days (for 3 cycles).
  Interventions: Drug: Erenumab-Aooe; Drug: Erenumab-Aooe Matching Placebo

INTERVENTIONS:
Drug: Siltuximab — A chimeric immunoglobulin G mAb, via intravenous infusion.
  Other Names: Sylvant
  Arms: Sub-study A: Siltuximab
Drug: Erenumab-Aooe — Human monoclonal antibody, single-dose prefilled SureClick® autoinjector, via subcutaneous injection.
  Other Names: Aimovig
  Arms: Sub-study B: Erenumab-Aooe
Drug: Siltuximab Matching Placebo — Dextrose 5% in water, via intravenous infusion.
  Other Names: Normal Saline
  Arms: Sub-study A: Siltuximab
Drug: Erenumab-Aooe Matching Placebo — 0.9% saline, 1 mL single-dose prefilled syringe, via subcutaneous injection.
  Other Names: Normal Saline
  Arms: Sub-study B: Erenumab-Aooe

SUMMARY:
This is a placebo-controlled, multi-arm phase II platform screening trial designed to test the safety, pain responses, and pharmacodynamic activity of multiple experimental therapies simultaneously in participants with moderate-to-severe pain due to schwannomatosis (SWN).

This Master Study is being conducted as a platform that may allow participants with pain associated with schwannomatosis to receive a novel intervention throughout this study. Embedded within the Master Study are individual drug sub-studies:

* Investigational Drug Sub-Study A: Siltuximab
* Investigation Drug Sub-Study B: Erenumab-Aooe

DETAILED DESCRIPTION:
This is a placebo-controlled, multi-arm phase II platform screening trial designed to test the safety, pain responses, and pharmacodynamic activity of multiple experimental therapies simultaneously in participants with moderate-to-severe pain due to schwannomatosis (SWN).

The MASTER STUDY has no study drug or intervention. It is intended to enroll participants who will be placed into different treatment arms (SUB-STUDIES), which will each have an additional consent and enrollment process.

MASTER STUDY

* The research study procedures include screening for eligibility, randomization to an experimental treatment sub-study, if qualified, and observation for up to 10 years.

  * Subjects who complete treatment on one experimental arm will be permitted to enroll in a different experimental treatment arm if they meet eligibility criteria.
  * Participants who are not eligible for enrollment in a different treatment sub-study will be permitted to remain under observation on this Master Study to understand the natural history of schwannomatosis-related pain and tumor growth pattern.
  * Participants will be eligible to remain on this Master Study for up to 10 years.
  * It is expected that about 40 people will take part in the Master Study.
  * The study will randomize a maximum of 20 participants to each of the experimental arms. The overall size of the trial is not fixed by design because it includes arm-dropping rules for futility and allow for the possibility of arm addition by amendment.
* Upon meeting Master Study qualifications, participant will be randomly assigned to a treatment sub-study.

SUB-STUDY A - SILTUXIMAB

* The purpose of this study is to find out what effects, good and/or bad, siltuximab has on schwannomatosis-associated pain.
* The U.S. Food and Drug Administration (FDA) has not approved Siltuximab for schwannomatosis but it has been approved for the treatment of people with multicentric Castleman's disease (MCD) who are human immunodeficiency virus (HIV) negative and human herpesvirus-8 (HHV-8) negative.
* Siltuximab was identified as a potential treatment for schwannomatosis tumors in a screen of compounds in a laboratory. Siltuximab is believed to work by blocking the growth signals and inflammation in tumor cells.
* Upon meeting sub-study qualifications, participant will be randomly assigned to either the early-start group or the delayed-start group.
* Twenty (20) people will take part in the siltuximab Sub-study.
* Participants in the early-start group will receive siltuximab every 3 weeks over 168 days. Participants in the delayed-start group will receive placebo every 3 weeks for the first 84 days followed by siltuximab every 3 weeks over the subsequent 84 days (for a total of 168 days).

SUB-STUDY B - ERENUMAB-AOOE

* The purpose of this study is to find out what effects, good and/or bad, erenumabaooe has on schwannomatosis-associated pain.
* The U.S. Food and Drug Administration (FDA) has not approved Erenumab-Aooe for schwannomatosis but has approved it for treatment of migraines headaches in adults.
* Erenumab-Aooe was identified as a potential treatment for schwannomatosis pain. Erenumab-aooe acts by blocking pain signals in the body. By blocking pain signals, erenumabaooe may reduce pain associated with schwannomatosis.
* Upon meeting sub-study qualifications, participant will be randomly assigned to either the early-start group or the delayed-start group.
* Twenty (20) people will take part in the ERENUMAB-AOOE Sub-study.
* Participants in the early-start group will receive erenumab-aooe every 4 weeks over 168 days. Participants in the delayed-start group will receive placebo every 4 weeks for the first 84 days followed by erenumab-aooe every 4 weeks over the subsequent 84 days (for a total of 168 days).

ELIGIBILITY:
Inclusion Criteria for Master Study:

* Patients must have a confirmed diagnosis schwannomatosis by fulfilling either clinical or molecular diagnosis.
* Clinical diagnosis: A clinical diagnosis of schwannomatosis is confirmed by either of the two following criteria:

  * Two or more non-intradermal schwannomas, one with pathological confirmation, without evidence of bilateral vestibular schwannoma (see exclusion criteria 3.2.3) OR
  * one pathologically confirmed schwannoma or intracranial meningioma and
  * An affected first-degree relative. Molecular diagnosis
* A molecular diagnosis of schwannomatosis is confirmed by either (1) two or more pathologically proven schwannomas or meningiomas AND genetic studies of at least two tumors with loss of heterozygosity (LOH) for chromosome 22 and two different NF2 mutations; or (2) one pathologically proven schwannoma or meningioma and a germline SMARCB1 or LZTR1 pathogenic mutation.
* Participant must be ≥ 18 years of age on Day 1 of treatment.
* Karnofsky performance status ≥ 70 or ECOG PS 0 or 1 (see Appendix A).
* Subject must have moderate-to-severe pain secondary to SWN, defined as Score ≥5 on the Numeric Rating Scale-11 (NRS-11) as the maximum pain intensity in the previous 7 days.
* Ability to understand and the willingness to sign written informed consent and assent documents.
* Must have established relationship with primary care physician and provide contact information.

Inclusion Criteria for Sub-study A - Siltuximab or Placebo Arm:

* Participants must be willing and able to provide written informed consent/assent for the siltuximab arm of the STARFISH trial.
* Subject must have moderate to severe pain secondary to schwannomatosis, defined as having a median Numeric Rating Scale-11 (NRS-11) score ≥5 during screening.
* Subject must have insufficient response to, intolerance of, be unwilling to try, or contraindication to medical therapies for SWN-related pain, such as NSAID therapy, opioid treatment, or neuropathic pain medications.
* Clinical laboratory values as specified below within 28 days before the first dose of study drug:

  * ALT/aspartate aminotransferase (AST) ≤ 2.5 × institutional upper limit of normal (ULN);
  * Total serum bilirubin ≤ 1.5 × institutional ULN (<3.0 × institutional ULN for patients with Gilbert syndrome)
  * Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2, using the modification of diet in renal disease (MDRD) equation
  * Serum lipase ≤1.5 × institutional ULN
  * Absolute neutrophil count ≥1.5 × 109/L
  * Platelet count ≥75 × 109/L
  * Hemoglobin ≥9 g/dL and <17 g/dL
* Female subjects of childbearing potential and at risk for pregnancy (e.g., not abstinent) must agree to use 2 highly effective methods of contraception throughout the study and for 100 days (15 weeks) after the last dose of assigned study medication.
* Female subjects of non-childbearing potential must meet at least 1 of the following criteria:

  * Have undergone documented total hysterectomy or bilateral oophorectomy
  * Have medically confirmed ovarian failure
  * Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; [status may be confirmed with/and have] a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state; In the event of indeterminate or anomalous results on pregnancy/FSH testing or issues surrounding contraceptive requirements, the study clinician should be contacted and will make the final decision as to the adequacy/need for contraception.

Inclusion Criteria for Sub-study B - Erenumab-Aooe or Placebo Arm:

* Participants must be willing and able to provide written informed consent/assent for the erenumab-aooe arm of the STARFISH trial.

  * Subject must have moderate to severe pain secondary to schwannomatosis, defined as a median NRS-11 Score ≥5 during Screening.
  * Subject must have insufficient response to, unwillingness to take, intolerance of, or contraindication to at least one medical therapies for SWN-related pain, such as NSAID therapy, opioid treatment, or neuropathic pain medications.
  * Clinical laboratory values as specified below within 28 days before the first dose of study drug:
* ALT/aspartate aminotransferase (AST) ≤ 2.5 × institutional upper limit of normal (ULN);
* Total serum bilirubin ≤ 1.5 × institutional ULN (<3.0 × institutional ULN for patients with Gilbert syndrome)
* Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2, using the modification of diet in renal disease (MDRD) equation
* Serum lipase ≤1.5 × institutional ULN
* Absolute neutrophil count ≥1.5 × 109/L
* Platelet count ≥75 × 109/L
* Hemoglobin ≥9 g/dL

  * Female subjects of childbearing potential and at risk for pregnancy (e.g., not abstinent) must agree to use 2 highly effective methods of contraception throughout the study and for 60 days after the last dose of assigned study medication.
  * Female subjects of non-childbearing potential must meet at least 1 of the following criteria:
* Have undergone documented total hysterectomy or bilateral oophorectomy
* Have medically confirmed ovarian failure
* Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; [status may be confirmed with/and have] a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state; In the event of indeterminate or anomalous results on pregnancy/FSH testing or issues surrounding contraceptive requirements, the study clinician should be contacted and will make the final decision as to the adequacy/need for contraception.

Exclusion Criteria for Master Study:

* Participants who have had chemotherapy within a minimum of 4 weeks prior to Master Study registration (or a minimum of 5 half-lives and resolution to baseline of toxicities unless there are irreversible toxicities from prior drug that do not influence risk of next drug).
* Participants who are receiving any other investigational agents.
* Participants with nervous system tumors that, in the opinion of the treating investigator, are likely to require active treatment (including surgery) within 6 months of registration to the Master Study.
* History of a malignancy in the last 3 years, unless (a) have been disease-free for at least 2 years or (b) are deemed by the treating investigator to be at low risk for progression or recurrence of that malignancy (e.g., carcinoma in situ, basal cell carcinoma, Gleason 6 prostate cancer) in the next 2 years
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Exclusion Criteria for Sub-study A - Siltuximab or Placebo Arm:

* Subject has a history of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG fusion protein.
* The subject's pain is related to a non-schwannomatosis cause such as prior cancer therapy, infection, bowel obstruction/perforation, spinal cord compression, or fracture or impending fracture of weight bearing bone.
* Subjects at increased risk for GI perforation including documented history of GI perforation, mesenteric ischemia, or intestinal volvulus; or chronic use of high dose glucocorticoids (particularly in combination with NSAIDs)
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Treatment with any investigational products within 1 month or 5 half-lives (whichever is longer) before the first dose of study drug
* Had major surgery within 30 days of the first dose of siltuximab. Minor surgical procedures such as catheter placement or minimally invasive biopsies are allowed.
* Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

  * Myocardial infarction within 6 months before the first dose of siltuximab.
  * Unstable angina within 6 months before first dose of siltuximab.
  * Congestive heart failure within 6 months before first dose of siltuximab.
  * History of clinically significant atrial arrhythmia (including clinically significant bradyarrhythmia), as determined by the treating physician.
  * Any history of clinically significant ventricular arrhythmia.
  * Had a cerebrovascular accident or transient ischemic attack within 6 months before first dose of siltuximab.
* Have uncontrolled hypertension (defined as an average systolic blood pressure > 160 or an average diastolic blood pressure > 100 for adults) despite adequate treatment with medications. Patients with hypertension should be under treatment on study entry to control blood pressure.
* Have an ongoing or active clinically significant infection, including, but not limited to, the requirement for intravenous antibiotics. Note: superficial infections that are treated with topical medications or other infections that, in the opinion of the site PI, are uncomplicated are not considered exclusion criteria.
* History of a malignancy in the last 3 years, unless (a) have been disease-free for at least 2 years or (b) are deemed by the treating investigator to be at low risk for progression or recurrence of that malignancy (e.g., carcinoma in situ, basal cell carcinoma, Gleason 6 prostate cancer) in the next 2 years.
* Have a known history of HIV infection. Testing is not required in the absence of history.
* Have any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of siltuximab.

Exclusion Criteria for Sub-study B - Erenumab-Aooe or Placebo Arm:

* Subject has a history of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG fusion protein
* Have chronic constipation limiting instrumental activities of daily living (e.g., laundry, dressing, shopping, running errands, and transportation).
* Have uncontrolled hypertension (defined as an average systolic blood pressure > 160 or an average diastolic blood pressure > 100) despite adequate treatment with medications. Patients with hypertension should be under treatment on study entry to control blood pressure
* The subject's pain is related to a non-schwannomatosis cause such as prior cancer therapy, infection, bowel obstruction/perforation, spinal cord compression, or fracture or impending fracture of weight bearing bone.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Treatment with any investigational products within 1 month or 5 half-lives (whichever is longer) before the first dose of study drug
* Had major surgery within 30 days of the first dose of erenumab-aooe. Minor surgical procedures such as catheter placement or minimally invasive biopsies are allowed.
* Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

  * Myocardial infarction within 6 months before the first dose of erenumab-aooe.
  * Unstable angina within 6 months before first dose of erenumab-aooe.
  * Congestive heart failure within 6 months before first dose of erenumab-aooe.
  * History of clinically significant atrial arrhythmia (including clinically significant bradyarrhythmia), as determined by the treating physician.
  * Any history of clinically significant ventricular arrhythmia.
  * Had a cerebrovascular accident or transient ischemic attack within 6 months before first dose of erenumab-aooe.
* History of a malignancy in the last 3 years, unless (a) have been disease-free for at least 2 years or (b) are deemed by the treating investigator to be at low risk for progression or recurrence of that malignancy (e.g., carcinoma in situ, basal cell carcinoma, Gleason 6 prostate cancer) in the next 2 years.
* Have a known history of HIV infection. Testing is not required in the absence of history.
* Have any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of erenumab-aooe.
* Participants who are lactating women are excluded from this study because there are no data on the presence of erenumab-aooe in human milk, the effects on the breastfed infant, or the effects on milk production.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in worst pain intensity for each drug sub-study | Baseline to week 12
  Defined as the change in the worst pain intensity between baseline and day 85. Worst pain is measured using the 11-point Pain Intensity Numerical Rating Scale (NRS), where scores range from 0 (no pain) to 10 (worst pain ever) of the maximum SWN-related pain experienced over the past week

SECONDARY OUTCOMES:
Number of Participants with Adverse Events in each drug sub-study | Randomization/1st treatment to 4 weeks post final treatment
  Graded according to NCI CTCAE v5.0. All participants will be evaluable for toxicity from the time of first treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Plotkin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Yin Z, Wu L, Zhang Y, Sun Y, Chen JW, Subudhi S, Ho W, Lee GY, Wang A, Gao X, Ren J, Zhu C, Zhang N, Ferraro GB, Muzikansky A, Zhang L, Stemmer-Rachamimov A, Mao J, Plotkin SR, Xu L. Co-Targeting IL-6 and EGFR signaling for the treatment of schwannomatosis and associated pain. bioRxiv [Preprint]. 2023 Feb 6:2023.02.06.527377. doi: 10.1101/2023.02.06.527377. PMID 36798353